CLINICAL TRIAL: NCT02696395
Title: RSA-measured in Vivo Migration and Micromotion in the DePuy Tri-lock, Corail and Deltamotion Hip Replacement Components: a Single-blinded Randomised Control Trial
Brief Title: RSA-measured in Vivo Migration and Micromotion in the DePuy Tri-Lock, Corail and Deltamotion Hip Replacement Components
Acronym: DePuy RSA RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DePuy RSA RCT
Record Dates: First submitted 2015-11-16; First posted 2016-03-02 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DePuy Tri-Lock® (Active Comparator): Total hip replacement with DePuy Tri-Lock® femoral stem and Deltamotion® acetabular component. The surgery will be conducted using a postero-lateral approach followed by post operative rehabilitation as per standard care.
  Interventions: Device: DePuy Tri-Lock® femoral stem + Deltamotion® acetabular component
- DePuy Corail® (Active Comparator): Total hip replacement with DePuy Corail® femoral stem and Deltamotion® acetabular component. The surgery will be conducted using a postero-lateral approach followed by post operative rehabilitation as per standard care.
  Interventions: Device: DePuy Corail® femoral stem + Deltamotion® acetabular component

INTERVENTIONS:
Device: DePuy Tri-Lock® femoral stem + Deltamotion® acetabular component
  Arms: DePuy Tri-Lock®
Device: DePuy Corail® femoral stem + Deltamotion® acetabular component
  Arms: DePuy Corail®

SUMMARY:
Hip replacements are being performed on an increasingly active population, who are likely to wear their implants out prematurely. New hip replacements have been devised to minimise the risk of failure. DePuy RSA RCT is a randomised controlled trial designed to compare the performance of two established types of hip replacements using Corail and Tri-Lock stems along with Deltamotion acetabular component. The primary objective of the trial is to compare the long term stability of these two devices.To do this, the study will use an advanced 3D Xray technique to detect migration of the components at 3 years. The study will also measure micromotion of Corail, Tri-Lock and Deltamotion components, patient reported outcome measures and change in bone density.This study is being conducted at a single site, at the Nuffield Orthopaedic Centre, Oxford.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 65 years and men aged between 18 and 70 years.

  * Participant is willing and able to give informed consent for participation in the study.
  * Diagnosed with hip osteoarthritis.
  * Able (in the Investigators opinion) and willing to comply with all study requirements.
  * Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* Any patients with an inflammatory arthropathy, osteoporosis or deformities of the proximal femur.

  * Patients who have significant co-morbidities that would make follow-up difficult or uncomfortable.
  * Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-07; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Mean total Radio Stereometric Analysis (RSA) measured migration of DePuy Tri-Lock® femoral stem vs DePuy Corail® femoral stem (mm/yr). | 3 years

SECONDARY OUTCOMES:
Dynamically Inducible Micromotion (DIMM) of DePuy Corail®, Tri-Lock® and Deltamotion® components (mm/yr). | 3 years
Radio Stereometric Analysis (RSA) measured migration of DePuy Deltamotion® acetabular component | 3 years
Change in Oxford Hip Score (OHS) at three years. | 3 years
Change in bone density using Dual Energy X-Ray Absorptiometry (DEXA) scan at 12 months. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Nuffield Orthopaedic Centre, Oxford, United Kingdom